CLINICAL TRIAL: NCT03161977
Title: The Effect of Mannitol on Intraoperative Serum Potassium in Patients Undergoing Craniotomy：an Observational Study
Brief Title: The Effect of Mannitol on the Serum Potassium During Craniotomy
Status: Completed | Type: Observational
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: XYFY-2017-011
Record Dates: First submitted 2017-05-11; First posted 2017-05-22 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-01

CONDITIONS: Mannitol Adverse Reaction; Hyperkalemia
MeSH Terms: conditions — Hyperkalemia | interventions — Mannitol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mannitol: Mannitol was intravenous infused within 15-20 mins when drilling skull
  Interventions: Other: Mannitol

INTERVENTIONS:
Other: Mannitol — Mannitol was intravenous infused within 15-20 mins when drilling skull

SUMMARY:
This is an observational study designed to research the effect of mannitol on the concentration of intraoperative serum potassium in patients undergoing craniotomy, and to guide the safe use of mannitol during craniotomy.

DETAILED DESCRIPTION:
Patients were assigned to receive 20% mannitol (1g/kg) solution administered intravenously 15-20 minutes at the time of drilling skull.The serum potassium was measured by arterial blood gas analysis before infusion (T0), infusion finished (T1), 15min (T2), 30min (T3), 60min (T4) and 120min (T5) after infusion.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 70
* American Society of Anesthesiologists physical status I to II
* liver and kidney function is normal
* preoperative concentration of serum potassium was from 3.5 to 5.5 mmol/L

Exclusion Criteria:

* history or presence of congestive heart failure (New York Heart Association class III to IV)
* history or presence of renal failure(diabetes insipidus, or syndrome of inappropriate antidiuretic hormone secretion)
* intraoperative blood transfusion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who are received craniotomy
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
the concentration of serum potassium | two hours within infusioning mannitol
  measured by arterial blood gas analysis

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
IPD will be available when this trial is finished and the article have been published

REFERENCES:
- [Background] Quentin C, Charbonneau S, Moumdjian R, Lallo A, Bouthilier A, Fournier-Gosselin MP, Bojanowski M, Ruel M, Sylvestre MP, Girard F. A comparison of two doses of mannitol on brain relaxation during supratentorial brain tumor craniotomy: a randomized trial. Anesth Analg. 2013 Apr;116(4):862-8. doi: 10.1213/ANE.0b013e318282dc70. Epub 2013 Jan 25. PMID 23354336
- [Background] Maas AI, Dearden M, Teasdale GM, Braakman R, Cohadon F, Iannotti F, Karimi A, Lapierre F, Murray G, Ohman J, Persson L, Servadei F, Stocchetti N, Unterberg A. EBIC-guidelines for management of severe head injury in adults. European Brain Injury Consortium. Acta Neurochir (Wien). 1997;139(4):286-94. doi: 10.1007/BF01808823. PMID 9202767
- [Background] The Brain Trauma Foundation. The American Association of Neurological Surgeons. The Joint Section on Neurotrauma and Critical Care. Initial management. J Neurotrauma. 2000 Jun-Jul;17(6-7):463-9. doi: 10.1089/neu.2000.17.463. PMID 10937888
- [Background] Fanous AA, Tick RC, Gu EY, Fenstermaker RA. Life-Threatening Mannitol-Induced Hyperkalemia in Neurosurgical Patients. World Neurosurg. 2016 Jul;91:672.e5-9. doi: 10.1016/j.wneu.2016.04.021. Epub 2016 Apr 13. PMID 27086258
- [Background] Better OS, Rubinstein I, Winaver JM, Knochel JP. Mannitol therapy revisited (1940-1997). Kidney Int. 1997 Oct;52(4):886-94. doi: 10.1038/ki.1997.409. No abstract available. PMID 9328926
- [Background] Palma L, Bruni G, Fiaschi AI, Mariottini A. Passage of mannitol into the brain around gliomas: a potential cause of rebound phenomenon. A study on 21 patients. J Neurosurg Sci. 2006 Sep;50(3):63-6. PMID 17019386
- [Background] Rozet I, Tontisirin N, Muangman S, Vavilala MS, Souter MJ, Lee LA, Kincaid MS, Britz GW, Lam AM. Effect of equiosmolar solutions of mannitol versus hypertonic saline on intraoperative brain relaxation and electrolyte balance. Anesthesiology. 2007 Nov;107(5):697-704. doi: 10.1097/01.anes.0000286980.92759.94. PMID 18073543
- [Background] Seto A, Murakami M, Fukuyama H, Niijima K, Aoyama K, Takenaka I, Kadoya T. Ventricular tachycardia caused by hyperkalemia after administration of hypertonic mannitol. Anesthesiology. 2000 Nov;93(5):1359-61. doi: 10.1097/00000542-200011000-00036. No abstract available. PMID 11046231
- [Background] WINTERS RW, SCAGLIONE PR, NAHAS GG, VEROSKY M. THE MECHANISM OF ACIDOSIS PRODUCED BY HYPEROSMOTIC INFUSIONS. J Clin Invest. 1964 Apr;43(4):647-58. doi: 10.1172/JCI104950. No abstract available. PMID 14149918
- [Background] Stewart PA. Modern quantitative acid-base chemistry. Can J Physiol Pharmacol. 1983 Dec;61(12):1444-61. doi: 10.1139/y83-207. PMID 6423247
- [Background] Manninen PH, Lam AM, Gelb AW, Brown SC. The effect of high-dose mannitol on serum and urine electrolytes and osmolality in neurosurgical patients. Can J Anaesth. 1987 Sep;34(5):442-6. doi: 10.1007/BF03014345. PMID 3117392
- [Background] Hirota K, Hara T, Hosoi S, Sasaki Y, Hara Y, Adachi T. Two cases of hyperkalemia after administration of hypertonic mannitol during craniotomy. J Anesth. 2005;19(1):75-7. doi: 10.1007/s00540-004-0270-4. PMID 15674521